CLINICAL TRIAL: NCT03545815
Title: Phase I Study to Evaluate Treatment of CRISPR-Cas9 Mediated PD-1 and TCR Gene-knocked Out Chimeric Antigen Receptor (CAR) T Cells in Patients With Mesothelin Positive Multiple Solid Tumors.
Brief Title: Study of CRISPR-Cas9 Mediated PD-1 and TCR Gene-knocked Out Mesothelin-directed CAR-T Cells in Patients With Mesothelin Positive Multiple Solid Tumors.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-028
Record Dates: First submitted 2018-05-23; First posted 2018-06-04 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Solid Tumor, Adult
Keywords: mesothelin, CRISPR-Cas9, PD-1, TCR
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-mesothelin CAR-T cells (Experimental): Patients receive mesothelin-directed CAR-T cells infusion with dose escalation will occur using a standard 3+3 dose escalation approach, beginning in dose level I with dose cohorts and rules for escalation and de- escalation.
  Patients receive anti-mesothelin-CAR T cells on day 0.
  Interventions: Biological: anti-mesothelin CAR-T cells

INTERVENTIONS:
Biological: anti-mesothelin CAR-T cells — Cells will be infused on day 0.

SUMMARY:
Multiple solid tumors have positive targets of mesothelin expressed on the surfaces of the tumor cells, we use the technique of CRISPR-Cas9 to knocked out the PD-1 and TCR of chimeric antigen receptor (CAR) T cells to effect the immuno-microenvironment around tumors.

DETAILED DESCRIPTION:
1. To evaluate the feasibility and safety of CRISPR-Cas9 mediated PD-1 and TCR gene-knocked out chimeric antigen receptor (CAR) T cells in patients with mesothelin positive multiple solid tumors.
2. To evaluate the duration of in vivo persistence of transferred CAR-T cells.
3. To observe and measure anti-tumor responses for patients with detectable mesothelin positive tumor lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed with mesothelin positive multiple solid tumors.
2. Failure of at least one prior standard of care chemotherapy for advanced stage disease.
3. Subjects must have measureable disease as defined by RECIST 1.1 criteria or modified RECIST criteria.
4. Patients > 18 years of age.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-3.
6. Life expectancy > 12 weeks.
7. Satisfactory organ and bone marrow function as defined by the following (of note, the minimal blood counts should be in the absence of transfusion or cytokine support):

   i. Absolute neutrophil count > 1,000/μl ii. Platelets >75,000/μl iii. Hemoglobin > 9 g/dL iv. Bilirubin < 2.0x the institutional normal upper limit unless secondary to bile duct obstruction by tumor v. Creatinine < 1.5x the institutional normal upper limit vi. Albumin ≥2 vii. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 5x the institutional normal upper limit viii. Cardiac ejection fraction of >55% as measured by resting echocardiogram, with no significant pericardial effusion.
8. Blood coagulation parameters: PT such that international normalized ratio (INR) is ≤ 1.5 and a PTT < 1.2 time the upper limit of normal unless the patient is therapeutically anti-coagulated for history of cancer-related thrombosis and has stable coagulation parameters.
9. Ability to understand and the willingness to provide written informed consent.
10. Male and Female subjects of reproductive potential agree to use approved contraceptive methods (e.g. birth control pills, barrier device, intrauterine device, abstinence) and abstain from other methods of conception during the study and for 6 months following the study cell infusion or proof of sterility.

Exclusion Criteria

1. Sarcomatoid MPM histology which is known in the literature to not express mesothelin; biphasic MPM is also excluded.
2. This refers to non-commercially approved investigational drugs different than those used in this protocol.Participated in any other trial in which receipt of an investigational study drug occurred within 28 days prior to enrollment and anticipated treatment with another investigational product while on study.
3. Anticipated need for systemic chemotherapy within 2 weeks before apheresis and infusion of CART-meso cells.
4. Active invasive cancer other than the one of the three cancers in this study. Patients with active non-invasive cancers (such as non-melanoma skin cancer, superficial cervical and bladder and prostate cancer with PSA level < 1.0) are not excluded.CART-meso in mesothelin expressing cancers
5. HIV, HCV, or HBV infections
6. Active autoimmune disease (including but not limited to: systemic lupus erythromatosis, Sjogren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, etc.) requiring immunosuppressive therapy within the past 4 weeks, with exception of thyroid replacement.
7. Patients with ongoing or active infection.
8. Planned concurrent treatment with systemic high dose corticosteroids. Patients may be on a stable low dose of steroids (<10mg equivalent of prednisone) for chronic respiratory conditions.
9. Patients requiring supplemental oxygen therapy.
10. Prior therapy with gene modified cells.
11. Previous experimental therapy with SS1 moiety, murine or chimeric antibodies (human and humanized antibodies are allowed).
12. History of allergy to murine proteins
13. History of allergy or hypersensitivity to study product excipients (human serum albumin, DMSO, and Dextran 40)
14. Any clinically significant pericardial effusion; CHF (NY Heart Association Grade II-IV) or cardiovascular condition that would preclude assessment of mesothelin induced pericarditis or that may worsen as a result of toxicities expected for this study. This determination will be made by a cardiologist.
15. Any clinically significant pleural or peritoneal effusion that cannot be drained with standard approaches. An indwelling drainage device placed prior to enrollment is acceptable.
16. Pregnant or breastfeeding women. Female study participants of reproductive potential must have a negative urine pregnancy test of enrollment. A serum pregnancy test will be performed within 2 weeks before infusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2020-10-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
study of related adverse events | 24 weeks
  Grade 3 signs/symptoms, toxicities and clinical

SECONDARY OUTCOMES:
clinical responses to anti-mesothelin cell infusions | 24 weeks
  Disease control rate(DCR)

CONTACTS AND LOCATIONS:
Locations (1):
- Biotherapeutic Department and Hematology Department of Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No